CLINICAL TRIAL: NCT04417647
Title: A Prospective, Randomized, Open-label, Controlled, Exploratory Trial to Investigate the Safety and Tolerability of Topically Administered VZ in Healthy Male Subjects With Artificial Dermal Wounds
Brief Title: G-Wound (VZ for Wound Treatment)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glock Health, Science and Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-Wound_01
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Wounds; Wound Heal
Keywords: Wound; Healing
MeSH Terms: conditions — Wounds and Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Proximal wound SoC treatment - Distal wound VZ application
  Interventions: Device: VZ powder (purified clinoptilolite); Procedure: Standard of care (SoC)
- Group 2 (Experimental): Distal wound SoC treatment - Proximal wound VZ application
  Interventions: Device: VZ powder (purified clinoptilolite); Procedure: Standard of care (SoC)

INTERVENTIONS:
Device: VZ powder (purified clinoptilolite) — VZ powder will be applied topically to the open surface of the verum treatment-assigned wound to cover the entire wound area. Following each VZ application, wounds will be protected by wound dressing (non-adhesive wound dressing (AdapticTM) and conventional protective Mepore® dressing).
Procedure: Standard of care (SoC) — wound cleansing (0.9% saline solution) and wound dressing (non-adhesive wound dressing (AdapticTM) and conventional protective Mepore® dressing) will be applied to the SoC-assigned wound.

SUMMARY:
This is a prospective, randomized, open-label, controlled, exploratory trial that aims to investigate the local skin tolerability of topically administered VZ and to evaluate efficacy and safety parameters associated with improved wound condition and healing

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects
2. Age 18-45 years at time of screening
3. Subjects are in good clinical and mental health as established by medical history and physical examination
4. Subject agrees to be compliant with study related visit and treatment schedule
5. Written informed consent

Exclusion Criteria:

1. Regular use of medications affecting the blood clotting process (e.g. aspirin or any other over-the-counter medicine or complimentary health product affecting the blood clotting process) or immunosuppressive drugs. Aspirin should not be taken in the 10 days prior to study participation or during the study
2. Use of topical (in the skin area of investigation) or systemic antibiotics within the last 4 weeks before study enrolment
3. History of cancer (except for non-melanoma skin cancer) within the previous 12 months or treatment with anticancer therapy (chemotherapy, immunotherapy, radiotherapy, hormone therapy for cancer treatment, targeted therapy or gene therapy) within 12 months before the first administration of investigational product or at any time during the study
4. Subjects with any known coagulation disorder
5. Subjects who have pigmented skin (Fitzpatrick Classification Level V - VI) due to an increased susceptibility to hypertrophic and keloid scarring
6. History of wound healing abnormalities or a medical condition that is known to be associated with abnormal wound healing
7. Chronic inflammatory dermatological disease
8. History of chronic autoimmune diseases such as, but not restricted to rheumatoid arthritis, inflammatory bowel disease, lupus erythematodes
9. Subjects diagnosed with Diabetes Type I or II
10. Lack of 2-point discrimination above 10 cm as assessed using an aesthesiometer
11. Tattoos, scars, burns, rashes or hyper- or hypopigmentation in the region of planned punch biopsy
12. Evidence of active infectious disease including HIV and hepatitis B or C
13. Current smoker (or any kind of nicotine consumption)
14. Known allergies to biopsy numbing medication, wound cleansing solution and wound dressing
15. Known hypersensitivity to aluminium and/or silicon
16. Allergy requiring medical treatment within the last 4 weeks prior to screening
17. Active infection or fever > 38°C within the last 7 days prior to randomization
18. Clinically relevant abnormalities in the laboratory testing, vital signs, ECG or physical examination
19. Alcohol abuse or a positive urine screen for drugs of abuse at screening
20. Participation in another clinical trial with an investigational day within the last 4 weeks before study participation
21. Employee at the study site, spouse/partner or relative of any study staff (e.g. investigator, sub-investigators, or study nurse) or relationship to the sponsor

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Local tolerability of IMD | 14 days
  Local tolerability of IMD assessed using erythema severity score: a scale from 0 - 4 (0 = no visible reaction, 1 = faint, minimal erythema, 2 = erhythema, 3 = erythema with induration of vesicles, 4 = severe erythema with induration, vesicles or bullae or pustules and/ulceration) with 0 being best and 4 being worst.

SECONDARY OUTCOMES:
Change in wound size | 14 days
  Change in wound size between baseline and End of Treatment (EoT) assessed by photographic analysis
Wound closure | 1 day
  Presence or absence of complete wound closure at End of Treatment (EoT) visit
Wound healing and condition | 14 days
  Wound healing and wound condition parameters assessed as a dichotomous outcome by the investigator
Histological evaluation | 2 days
  Descriptive histological evaluation of wound healing by H&E and Masson trichrome staining as well as by immunostaining against biomarkers of the biopsy specimens obtained at baseline and at EoT
Investigator's satisfaction on topical applicability | 14 days
  Investigator's satisfaction on topical applicability of VZ evaluated via a 5-point Likert scale: a scale from 1 - 5: 5 = extremely satisfied, 4 = very satisfied, 3 = moderately satisfied, 2 = slightly satisfied, 1 = not at all satisfied) with 5 being best and 1 being worst.
Change in local pain intensity | 14 days
  Change in local pain intensity based on the Visual Analogue Scale (VAS) when compared to SoC-treated wounds with a scale from 0-10: 0 - no pain and 10 - worst possible pain.
Adverse Events and Serious Adverse Events | 28 days
  Incidence of treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, Prof.Dr., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No